CLINICAL TRIAL: NCT04817397
Title: The Lymphocyte/Neutrophil Ratio as a Prognostic Index for Short Term Outcome in the ICU Admitted COVID-19 Adult Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Professor Emad Zarief kamel, Assiut University
Other Study IDs: ICU admitted COVID-19 patients
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. ry outcome includes the correlation between lymphocyre /neurtophll ratio (LNR) and mortality rate during hospital stay in the ICU admitted COVID 19 patients.
2. ry outcome(s) include the LNR and its correlation with ICU stay, the need for mechanical ventilation, renal impairment.

DETAILED DESCRIPTION:
In December 2019,the COVID-19 virus has been mainly breaking out in Wuhan in China as pneumonia affecting patients . Common clinical features During hospitalization started to appear including acute respiratory infection , inflammatory reaction , fever, pneumonia, cough, fatigue , anosmia .

The patient known suspected if he has a clinical picture of viral pneumonia, exposure history, and radiographic findings [CT] or [MRI] chest consistent with COVID-19 pneumonia. the gold standard and the Final diagnosis (PCR) positivity for the presence of coronavirus .

The immune response to respiratory infection causes neutrophils to collect inside the lung especially the alveoli. Neutrophils aggregation may lead to collateral tissue damage and cytotoxicity. According to Previous studies apoptosis of lymphocytes occurred due to the release of anti-inflammatory cytokines resulting in lymphopenia. high levels of circulating neutrophils have been demonstrated in COVID-19 patients(

A lot of literatures and studies have demonstrated the value of what is called neutrophil/ lymphocyte ratio (LNR) as a simple prognostic ratio correlated to morbidity and mortality. Up to our knowledge, there is no study utilized such ratio in COVID-19 ICU admitted patients, so that, this study has been built

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged ≥18 years)
2. Patients who need non-invasive ventilation (NIV or CPAP) or invasive ventilation (intubation)

Exclusion Criteria:

1. Previous diagnosis of severe liver or kidney failure.
2. Patients with Human Immunodeficiency Virus (HIV) infection.
3. Patients with previous hematological diseases (Leukemia) that condition alterations in blood counts.
4. Consumption of treatments with any type of immunosuppressants prior to admission that conditions low lymphocytes.
5. Patients with bone marrow depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will conducted on admitted patients that diagnosed as COVID at Assiut university hospitals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
The Lymphocyte/neutrophil ratio | up to 30 days
  The Lymphocyte/neutrophil ratio as a prognostic index for short term outcome in the ICU admitted COVID-19 adult patients

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit University, Asyut, Egypt

REFERENCES:
- See also: NEUTROPHIL TO LYMPHOCYTE RATIO VS PLATELETS TO LYMPHOCYTE RATIO: BIOMARKERS TO PREDICT SEVERITY OF DISEASE AND THEIR COMPARISON IN PATIENTS OF COVID-19 — https://pafmj.org/index.php/PAFMJ/article/view/5010